CLINICAL TRIAL: NCT02765178
Title: Apathy in Tourette Syndrome and Changes in Quality of Life - Effect of Medications
Brief Title: Apathy in Tourette Syndrome and Changes in Quality of Life
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201500989
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Tourette Syndrome; Apathy
MeSH Terms: conditions — Tourette Syndrome; Lethargy | interventions — Demography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Tourette Syndrome: The primary caregiver will be asked to fill the Children's motivation Scale. Other measures will be collected including a clinician filled Yale Global Tic Severity Scale (YGTSS) - severity score, Center for Epidemiological Studies Depression Scale for Children (CES-DC) and Gilles de la Tourette Syndrome Quality Of Life scale (GTS-QOL). Demographic data will also be collected for each study patient. Demographic data will also be collected for each study patient.
  Interventions: Other: Children's Motivation Scale; Other: Yale Global Tic Severity Scale (YGTSS); Other: Studies Depression Scale for Children (CES-DC); Other: Gilles de la Tourette Syndrome Quality Of Life scale; Other: Demographic Data
- Patients with Diabetes type 1: The primary caregiver will be asked to fill the Children's motivation Scale. Demographic data will also be collected for each study patient.
  Interventions: Other: Children's Motivation Scale

INTERVENTIONS:
Other: Children's Motivation Scale — A 16-item questionnaire to evaluate level of motivation in children and adolescents completed by the primary caregiver.
Other: Yale Global Tic Severity Scale (YGTSS) — Clinician administered questionnaire given to Tourette patients. Part 1 asks about 10 types of motor tics, 12 types of vocal tics (current, ever, age of onset, description). Part 2 is a severity rating that scores both motor and vocal tics on a 0-5 scale for each severity item: number of tics, intensity, frequency, complexity, interference, impairment. Totals are summed for all items.
  Groups: Patients with Tourette Syndrome
Other: Studies Depression Scale for Children (CES-DC) — Clinician administered questionnaire given to Tourette patients. Consisting of 20 items, respondents are asked to indicate how strongly they have felt a certain way during the past week using a Likert-type scale that ranges from "not at all" to "a lot." Only two items on the questionnaire relate specifically to sleep or fatigue. CES-DC is a validated score for assessing depression in children and adolescents
  Groups: Patients with Tourette Syndrome
Other: Gilles de la Tourette Syndrome Quality Of Life scale — Clinician administered questionnaire given to Tourette patients. Gilles de la Tourette Syndrome Quality Of Life scale (GTS-QOL) is a recently validated score for the assessment of quality of life in patients with Tourette syndrome. Consisting of a 27-item GTS-specific HR-QOL scale (GTS-QOL) with four subscales (psychological, physical, obsessional, and cognitive).
  Groups: Patients with Tourette Syndrome
Other: Demographic Data — Data will be collected including: age, age at disease onset, gender, current medication regimen and presence of co-morbidities (like a diagnosis of ADHD, OCD, depression or insomnia).
  Groups: Patients with Tourette Syndrome

SUMMARY:
Tourette syndrome is a complex neuropsychological disorder with both motor and vocal tics associated with multiple psychological co-morbidities. Apathy has not been widely studied in patients with Tourette syndrome. Apathy can result in decrease in self-care and disease control. In this study investigators will compare the occurrence of apathy in the adolescent Tourette syndrome population (at the UF center for movement disorders and Neurorestoration) to an age and gender matched control population. Investigators will also assess the role of commonly used medications in the Tourette population (neuroleptics and selective serotonin receptor inhibitors) in the occurrence of apathy.

DETAILED DESCRIPTION:
Tourette syndrome(TS) is a complex neuropsychological disorder with both motor and vocal tics associated with multiple psychological co-morbidities. The most common co-morbidities include obsessive compulsive disorder (OCD), attention deficit and hyperactivity disorder (ADHD) and depression. Apathy has not been extensively studied in the Tourette syndrome population. Apathy is currently defined as reduced motivation, with symptoms in at least two of three domains of reduced initiative, reduced interest and/or reduced emotional responsiveness. A study assessed the prevalence of apathy in multiple movement disorders and reported that apathy is much more common in disorders associated with slowed movements like Parkinson disease while less common in disorders with increased movements like Huntington disease and Tourette syndrome in adults. However, no apathy studies in adolescent patients with Tourette syndrome are published. Disengagement from treatment may affect health outcomes in other disease states. Apathy has significant effects on the quality of life and health outcomes in many patients. Apathy can be a direct manifestation of the neuropsychological process (intrinsic to the disease) or can be secondary to medication side effects most notably anti-dopaminergic agents and some reports of selective serotonin receptor inhibitors (SSRI). Further attention to the prevalence and impact of apathy in the adolescent Tourette syndrome population is needed to explore if this may be a factor influencing TS management and ultimately Quality of life (QOL). Multiple psychotropic medications are used in the management of tics as well as the psychological co-morbidities. How these medications affect apathy prevalence in Tourette syndrome patients is not known.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Tourette syndrome
* Age: 12-16 years
* Followed at the CMDNR

Exclusion Criteria:

* History of cerebral palsy or traumatic brain injury

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Targeted study population includes patients 12-16 years old diagnosed with Tourette Syndrome who are a patient of University of Florida Movement Disorders Center.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Children's Motivation Scale | Day 1
  A 16-item questionnaire to evaluate level of motivation in children and adolescents completed by the primary caregiver.

SECONDARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | Day 1
  Clinician administered questionnaire given to Tourette patients. Part 1 asks about 10 types of motor tics, 12 types of vocal tics (current, ever, age of onset, description). Part 2 is a severity rating that scores both motor and vocal tics on a 0-5 scale for each severity item: number of tics, intensity, frequency, complexity, interference, impairment. Totals are summed for all items.
Studies Depression Scale for Children (CES-DC) | Day 1
  Clinician administered questionnaire given to Tourette patients. Consisting of 20 items, respondents are asked to indicate how strongly they have felt a certain way during the past week using a Likert-type scale that ranges from "not at all" to "a lot." Only two items on the questionnaire relate specifically to sleep or fatigue. CES-DC is a validated score for assessing depression in children and adolescents
Gilles de la Tourette Syndrome Quality Of Life scale | Day 1
  Clinician administered questionnaire given to Tourette patients. Gilles de la Tourette Syndrome Quality Of Life scale (GTS-QOL) is a recently validated score for the assessment of quality of life in patients with Tourette syndrome. Consisting of a 27-item GTS-specific HR-QOL scale (GTS-QOL) with four subscales (psychological, physical, obsessional, and cognitive).

CONTACTS AND LOCATIONS:
Overall Officials: Wissam Deeb, Principal Investigator — UF Center for Movement Disorders and Neurorestoration
Locations (1):
- UF Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No